CLINICAL TRIAL: NCT04291807
Title: Determining the Effect of Video Assisted Education on Anxiety Level and Satisfaction Before ERCP Procedure
Brief Title: Video Assisted Education Before ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, leylacevik, Research Nurse, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERCPvideo
Record Dates: First submitted 2020-02-13; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Patient Compliance
Keywords: video education; ERCP; anxiety level; pain score
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video education (Experimental): A video of ERCP procedure has been viewed to the patients who will undergo ERCP and questions about the procedure had been answered by the primary investigator (experienced endoscopy nurse)
  Interventions: Behavioral: Video education
- Direct ERCP (No Intervention): Patients arranged ERCP for any reason underwent directly to the ERCP without any video education.

INTERVENTIONS:
Behavioral: Video education — Procedure was presented to the cases via a video showing the steps in ERCP and questions had been answered by an experienced nurse
  Arms: Video education

SUMMARY:
It was aimed to study the effect of video assisted education about endoscopic retrograde cholangiopancreaticography (ERCP) on anxiety levels of patients who planned to undergo ERCP for any reason.Video revealing the ERCP procedure was shown to the patients in one group and not shown to the other. Then anxiety levels and pain scores have been obtained before and after the procedure in both groups

DETAILED DESCRIPTION:
The study was conducted to determine the effect of video education on anxiety level before the ERCP procedure and satisfaction degree after the ERCP procedure between September 1st 2017 and December 31st 2018 at Bagcilar Medipol Mega University Hospital. Patients were grouped into two in a randomized manner. In control arm, patients underwent ERCP procedure with the information provided by the gastroenterologist who recommended the procedure. Patients in experimental arm, besides the information provided by the gastroenterologist, watched video of ERCP procedure and answered all the questions about the procedure by an experienced nurse. A total of 70 patients (35 in each arms) was planned to enroll to the study. State-Trait Anxiety Inventory (STAI) form was applied to measure anxiety level and visual analog score (VAS) was applied to measure the satisfaction about the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Conscious enough to understand the procedure and education
* Patients who can read
* Hemodynamically stable patients
* Mentally stable patients
* Patients who gave informed consent

Exclusion Criteria:

* Patients who underwent previous ERCP procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Change in anxiety status of the patients after ERCP | an hour before ERCP and an hour after ERCP
  This will be measured with Stait Trait Anxiety Inventory. There are 2 subscales within this measure. The State Anxiety Scale (S-Anxiety) evaluates the current state of anxiety, asking how respondents feel "right now," using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system. The Trait Anxiety Scale (T-Anxiety) evaluates relatively stable aspects of "anxiety proneness," including general states of calmness, confidence, and security.
  The STAI has 40 items, 20 items allocated to each of the subscales. Responses for the S-Anxiety scale assess intensity of current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Responses for the T-Anxiety scale assess frequency of feelings "in general": 1) almost never, 2) sometimes, 3) often, and 4) almost always.
  Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.

SECONDARY OUTCOMES:
Satisfaction assessed by visual analogue scale | an hour after ERCP
  A VAS for satisfaction is a horizontal line of 100-mm long. At the beginning and at the end, there are two descriptors representing extremes of satisfaction (i.e. no satisfaction and extreme satisfaction). The patient rated his satisfaction by making a vertical mark on the 100-mm line. The measurement in millimetres was converted to the same number of points ranging from 0 to 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Cevik, RN, Principal Investigator — Medipol University; Selda Rızalar, Assoc Prof, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No